CLINICAL TRIAL: NCT07064564
Title: A Randomized, Active-comparator Controlled, Two-Dose-level Study of iSTEP-N in Healthy Adults With Long Term Safety and PK Follow-up
Brief Title: iSTEP-N 101b: Pharmacokinetics and Safety Study of Low- and High-Dose Naltrexone Implants vs Monthly Vivitrol in Healthy Volunteers
Acronym: iSTEP-N
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akyso Therapeutics, LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Cenexel JBR (Unknown); Fast-Track Drugs & Biologics, LLC (Unknown); Aliri Bioanalysis (Unknown); Ardena (Unknown); Element Analytics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iSTEP-N 101b; UH3DA048338 (NIH)
Record Dates: First submitted 2025-07-05; First posted 2025-07-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Opioid Use Disorder
Keywords: naltrexone; biopin; oud; implant; opioid use disorder; extended-release; vivtrol
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of three parallel groups: (1) low-dose iSTEP-N implant, (2) high-dose iSTEP-N implant, or (3) monthly Vivitrol injections. All groups are followed concurrently for 12 months to assess pharmacokinetics and safety. Participants who receive an iSTEP-N implant may continue in a longer-term follow-up phase to evaluate implant persistence and extended pharmacokinetics.
Masking Description: This is an open-label study. No masking is used due to the differences in route of administration between the implant and injectable comparator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- iSTEP-N High Dose Implant (Experimental): Participants in this arm will receive a single subcutaneous implant of iSTEP-N at a high dose level (14.4 grams of naltrexone) on Day 1. Participants will undergo pharmacokinetic and safety evaluations for 12 months. Participants with a detectable implant or measurable naltrexone levels at the end of this period may continue in a longer-term follow-up phase.
  Intervention:
  Drug: iSTEP-N Naltrexone Implant - High Dose Single 14.4 g subcutaneous implant administered on Day 1.
  Interventions: Drug: Naltrexone implant, 14.4 grams
- Low-Dose iSTEP-N Implant (Experimental): Arm Description (Revised - Low-Dose iSTEP-N) Participants in this arm will receive a single subcutaneous implant of iSTEP-N containing 9.6 grams of naltrexone on Day 1. Participants will undergo pharmacokinetic and safety evaluations for 12 months. Participants with a detectable implant or measurable naltrexone levels at the end of this period may continue in a longer-term follow-up phase.
  Intervention:
  Drug: iSTEP-N Naltrexone Implant (Low Dose) Single 9.6 g subcutaneous implant administered on Day 1.
  Interventions: Drug: Naltrexone implant, 9.6 grams
- Vivitrol Injection (Active Comparator): Participants in this arm will receive 380 mg of extended-release naltrexone (Vivitrol) by intramuscular injection every 4 weeks for 12 months. Blood samples will be collected to evaluate pharmacokinetics and safety.
  Intervention:
  Drug: Vivitrol (Extended-Release Naltrexone Injection) 380 mg IM injection every 4 weeks for 52 weeks.
  Interventions: Drug: Extended-release naltrexone injection, 380 mg

INTERVENTIONS:
Drug: Naltrexone implant, 14.4 grams — Subcutaneous bioresorbable implant containing 14.4 grams of naltrexone, inserted into the thigh on Day 1 and designed to release drug steadily over 12 months.
  Arms: iSTEP-N High Dose Implant
Drug: Naltrexone implant, 9.6 grams — Subcutaneous bioresorbable implant containing 9.6 grams of naltrexone, inserted into the thigh on Day 1 and designed to release drug steadily over 12 months.
  Arms: Low-Dose iSTEP-N Implant
Drug: Extended-release naltrexone injection, 380 mg — Intramuscular injection of 380 mg extended-release naltrexone (Vivitrol), administered every 4 weeks for 12 months as the active comparator.
  Arms: Vivitrol Injection

SUMMARY:
This Phase 1b clinical study is evaluating iSTEP-N, an investigational extended-release implant containing naltrexone, a medication used to block the effects of opioids. The implant is placed under the skin of the thigh and is designed to release medication continuously over many months.

The main purpose of the study is to measure blood levels of naltrexone over time after administration of two different doses of the iSTEP-N implant and to compare those levels with the blood levels achieved by Vivitrol®, an FDA-approved injectable extended-release naltrexone given once every month.

The study will enroll healthy adult volunteers aged 18 to 65 years. Participants will be randomly assigned to one of three groups:

* Low-dose iSTEP-N implant
* High-dose iSTEP-N implant
* Monthly Vivitrol injections

Participants will be followed closely for approximately 12 months to measure medication levels and monitor safety, side effects, and overall health. The study will help determine whether the iSTEP-N implant can maintain naltrexone levels comparable to or higher than those achieved with monthly injections, especially during periods when protection from relapse is most important.

Participants who receive an iSTEP-N implant and still have detectable implant material or measurable medication levels at the end of the first year may continue in a long-term follow-up period lasting up to two additional years. During this period, researchers will monitor how long the implant remains detectable and how long medication continues to be released. If the implant remains after two years, participants may choose to have it surgically removed or simply end study participation.

The study is sponsored by Akyso Therapeutics, LLC, with clinical operations conducted at a dedicated clinical research center and oversight provided by an independent Institutional Review Board. All participants undergo screening examinations to confirm eligibility and are carefully monitored throughout participation.

Results from this study will help determine the appropriate dose of iSTEP-N for future clinical trials and support development of long-acting treatment options for opioid use disorder that may reduce the need for frequent injections.

DETAILED DESCRIPTION:
Opioid use disorder (OUD) remains a major public health challenge, driven in part by relapse and overdose risk after detoxification. Extended-release naltrexone, an opioid receptor antagonist, is approved as a once-monthly intramuscular injection (Vivitrol®) and reduces relapse risk by blocking opioid effects. However, treatment adherence may be limited by the need for repeated clinic visits and injections, and drug levels decline toward the end of each dosing interval, potentially reducing protection during periods of highest relapse vulnerability.

iSTEP-N is an investigational subcutaneous implant designed to provide long-term delivery of naltrexone from a biodegradable polymer matrix. After placement beneath the skin of the thigh, the implant slowly releases medication over many months and gradually resorbs. Sustained medication delivery may improve adherence compared with monthly injections and maintain opioid receptor blockade without requiring repeated dosing visits.

Protocol iSTEP-N 101b is a Phase 1b study in healthy volunteers designed to further characterize pharmacokinetics and safety of extended-release naltrexone delivered via iSTEP-N implants compared with monthly injectable naltrexone. The study evaluates two implant dose levels in parallel with active-comparator treatment to determine whether the implant can maintain plasma naltrexone concentrations comparable to or exceeding those achieved with monthly injections over a one-year period.

The primary focus of the study is characterization of plasma concentrations of naltrexone over time and estimation of pharmacokinetic parameters that describe drug exposure following implant placement. Secondary analyses include evaluation of concentrations of the major metabolite, 6β-naltrexol, and assessment of safety and tolerability across treatment groups.

Because the investigational product is a drug-device combination, the protocol also evaluates implant site outcomes and the duration of implant detectability and drug release. Participants receiving iSTEP-N who continue to have detectable implant material or measurable naltrexone levels after the first year may enter a long-term follow-up phase. This phase allows investigators to determine how long the implant continues to release drug and when the implant is no longer detectable by clinical examination or imaging.

The study design incorporates staged enrollment and independent safety monitoring to ensure early identification of any safety concerns during implant administration and follow-up. Frequent safety assessments are performed throughout participation, including monitoring for implant site reactions and systemic adverse effects associated with naltrexone.

Results from this study are intended to guide dose selection and study design for subsequent clinical development of long-acting naltrexone implants aimed at reducing barriers to sustained opioid relapse prevention therapy.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for the study:

Healthy adult male or female volunteers, ages 18 to 55 years.

Able and willing to provide written informed consent prior to any study procedures.

In good general health as determined by medical history, physical examination, vital signs, ECG, and laboratory tests (chemistry, hematology, and coagulation).

No clinically significant abnormalities in lab results, as determined by the investigator.

Negative urine drug screen for opioids, cocaine, amphetamines, benzodiazepines, cannabinoids, and other substances of abuse.

Negative breath alcohol test at screening and baseline.

Negative naloxone challenge test, indicating no physiological opioid dependence.

For females of childbearing potential:

Negative serum pregnancy test at screening and Day 0.

Agreement to use acceptable contraception (including oral hormonal contraception) for the duration of the study.

For males with female partners of childbearing potential:

Agreement to use effective contraception throughout the study.

Negative infectious disease panel, including HIV, hepatitis B surface antigen, and hepatitis C antibody.

No evidence of suicidal ideation or behavior on the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening.

Hamilton Depression Rating Scale (HAM-D17) total score of 0 to 10, consistent with no or minimal depressive symptoms.

Willing and able to comply with all study visits, procedures, and restrictions, including pharmacokinetic sampling.

Willing to refrain from donating blood during the study period.

Agree not to use opioid-containing medications for the duration of the study unless medically necessary and approved by the investigator.

Exclusion Criteria:

Participants who meet any of the following conditions will be excluded:

Current or recent history (past 12 months) of opioid use disorder, substance use disorder, or alcohol dependence.

Positive urine drug test or breath alcohol test at screening or prior to randomization.

Failure of the naloxone challenge test, indicating possible physical opioid dependence.

Use of any investigational drug or device within 30 days prior to screening.

Use of any opioid-containing medications (prescription or OTC) within 14 days prior to screening.

Known hypersensitivity or allergy to naltrexone, polycaprolactone (PCL), polylactic acid (PLA), polymeric implants, or any other component of the study drug.

History of chronic pain, neurological or psychiatric disorders, or any condition requiring regular use of medications.

Active medical condition or past medical history that, in the opinion of the investigator, could interfere with the study or pose an undue risk, including:

Cardiovascular disease

Hepatic or renal impairment

Gastrointestinal disorders affecting absorption

Respiratory disease

Seizure disorder

Autoimmune or inflammatory disorders

Females who are pregnant, breastfeeding, or planning to become pregnant during the study period.

Baseline systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg.

History of major depressive disorder, bipolar disorder, psychosis, or other severe psychiatric illness.

HAM-D17 score >10 at screening or Day 0.

Any suicidal ideation or behavior as defined by the C-SSRS in the past 6 months.

Participation in another clinical trial with investigational medication or device within the past 30 days.

Known coagulation disorder or current use of anticoagulants.

Inability to comply with study procedures due to geographic, social, or mental limitations.

Presence of any implantable medical device that may interfere with study procedures or assessments.

History of keloid formation or abnormal wound healing, which may affect implant insertion site.

History of HIV, hepatitis B, or hepatitis C, unless determined to be false positive or clinically insignificant by the investigator.

Any condition that, in the investigator's opinion, would make the subject unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Average plasma naltrexone concentration on the last day of each 4-week interval through Week 52 | Day 28, 56, 84, 112, 140, 168, 196, 224, 252, 280, 308, and 336
  The average of plasma naltrexone concentrations measured on the final day of each 4-week period through 12 months. This composite measure is used to assess sustained drug exposure and compare treatment arms.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) for Naltrexone | Day 1 through Week 52
  Total systemic exposure to naltrexone, calculated using AUCt and AUC∞ over the full study duration.
Maximum plasma concentration (Cmax) of naltrexone | Day 1 through Week 52
  Peak concentration observed post-dosing, determined by serial pharmacokinetic sampling.
Minimum plasma concentration (Cmin) of naltrexone | Day 1 through Week 52
  Lowest concentration between dosing intervals, providing information on potential trough levels.
Plasma concentration of 6β-naltrexol (naltrexone metabolite) | Day 1 through Week 52
  Metabolite levels measured alongside naltrexone to assess metabolism and systemic exposure.
Number of participants with treatment-emergent adverse events | Day 1 through Week 52
  Number of subjects experiencing adverse events related to study drug or procedures, including local and systemic findings.
Change in HAM-D17 depression scores from baseline | Baseline, Week 2, Week 4, and Week 24
  The Hamilton Depression Rating Scale-17 Item (HAM-D17) is a clinician-administered measure of depressive symptoms. Scores range from 0 to 52, with higher scores indicating more severe depression (worse outcome). Change from baseline will be assessed to monitor for worsening depressive symptoms or emergence of suicidality.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, Principal Investigator — MD

IPD SHARING:
Plan to Share IPD: No
This is a Phase 1b study in healthy volunteers designed to evaluate pharmacokinetics and safety of an investigational implant. Individual participant data (IPD) will not be shared because the study is not powered for clinical outcomes, involves no therapeutic intervention, and is not intended to support a comparative treatment analysis. Summary results will be reported in accordance with ClinicalTrials.gov requirements.